CLINICAL TRIAL: NCT03950375
Title: Round Window Visibility Prediction From Preoperative Scanner in Cochlear Implantation: Literature Review and Radiologic Criteria Evaluation
Brief Title: Radiologic Criteria for Round Window Visibility Prediction in Cochlear Implantation
Acronym: R-PO18155
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18155
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cochlear Implantation
Keywords: Sensorineural Hearing Loss; Round Window; ear surgery; Cochlear implantation
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cochlear implantation: "cochlear implantation" group : patients undergoing cochlear implantation between December 2018 and June 2019 in the ENT service of Reims universitary hospital.

SUMMARY:
The aim of the study is to identify the scannographic criterion the most relevant to predict the round window visibility during cochlear implantation.

DETAILED DESCRIPTION:
Whereas several surgical techniques exist to perform a cochlear implantation, the most used is the realization of mastoidectomy followed by posterior tympanotomy, in order to expose the round window, which finally permits to access to the cochlea. This procedure might be complicated with facial paresis, loss of residual hearing, because of anatomy relationships in this millimetric area.

CT scan of temporal bone is part of systematic preoperative assessment. Technological advances in radiology during the last decades now provide inframillimetric resolution. Thus, otologic surgeons wish they could anticipate round window exposure from these CT scan. This could decrease the procedure duration, complication occurrence, or improve surgical strategy.

Several studies proposed radiological criteria in this aim, from more or less complex measures in preoperative temporal bone CT scan. However, these diagnostic tests performances have not been assessed for most of them, or compared between them.

ELIGIBILITY:
inclusion criteria :

* patients undergoing cochlear implantation in Reims universitary hospital during the inclusion period
* patients who agree to participate in the study
* patients who had preoperative temporal bone CT scan

exclusion criteria : patients who have :

* temporal bone malformation on temporal bone CT scan or MRI
* chronic otitis media (except simple middle ear effusion)
* middle ear surgery antecedent
* cochlear implant in the context of a reimplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cochlear implantation
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
peroperative round window exposure | Day 0
  peroperative round window exposure evaluated according to St Thomas' Hospital classification:
  * visible (classes I and II) and not visible (class III)
  * easily visible (classes I and IIa) and not easily visible (class IIb and III)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France